CLINICAL TRIAL: NCT00738283
Title: Zinc and Copper Absorption in Neonates With Bilious Losses
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Steve Abrams, MD, Professor, Baylor College of Medicine
Other Study IDs: H-23224
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Ileostomy
Keywords: Zinc; Copper; Neonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, stool, gastric residuals, and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose to examine the absorption and excretion of zinc and copper in infants with ostomies. This will be accomplished by measuring baseline excretion and serum levels of zinc, copper, and ceruloplasmin, and by utilizing stable isotopes of zinc and copper to measure absorption and excretion.

To determine how the presence of an ileostomy impacts zinc and copper metabolism in infants at three time points: 1) when the infant has an ostomy and is receiving the majority of calories from total parenteral nutrition (TPN); 2) when the infant has an ostomy and is receiving primarily enteral nutrition without TPN; and 3) when/if the infant has a surgery to reconnect the bowel and is receiving primarily enteral nutrition.

For the first part of the study, excretion data for zinc will be obtained for ostomy patients. We hypothesize that infants with an ostomy will excrete more zinc in their stools than healthy term or preterm infants without ostomies.

For the second part of the study, we will obtain data on zinc absorption, secretion, and excretion through use of stable isotopes. Jalla et al determined that healthy infants retain zinc of 0.4 mg/day. We hypothesize that due to increased zinc losses, the infants in the study will be less positive than the healthy infants in the study by Jalla et al. Our study is designed to be able to detect if the ostomy patients net retention is one-half that described by Jalla (i.e. 0.2 mg/d). We will also obtain data on copper absorption, secretion, and excretion through the use of stable isotopes in the second part of the study. As a pilot study, we do not fully know what to expect regarding copper levels in infants with ostomies, but we hypothesize that they may be less positive than healthy infants without ostomies. Also, we hypothesize that zinc and copper are competitively absorbed in the gut; therefore, infants who receive more zinc may absorb less copper.

For the third part of the study, we will obtain data on zinc absorption through the use of stable isotopes after the infant has had surgery to reanastomose the bowel. We hypothesize that there may be continued zinc losses above those documented for healthy infants who have never had an ostomy, but decreased losses compared to when the infant had an ostomy.

DETAILED DESCRIPTION:
Potential subjects will be identified by study personnel in the Neonatal Intensive Care Units (NICU) of Texas Children's Hospital and Ben Taub General Hospital. The parent/guardian will be approached and the study will be explained in full. A time for questions will be allowed. Once the parent/guardian agrees to his/her child's participation, an informed written consent form will be signed. Subject confidentiality will be maintained within the limits of the law. All names and personal information will be accessed only by the investigators and authorized personnel. There will be no possibility of coercion as subjects will not have any relationship of dependency with the investigators.

We intend to asses zinc and copper metabolism at three time points: first, when the infant has an ostomy and is receiving primarily intravenous nutrition, called total parenteral nutrition (TPN), with minimal or no enteral feeds (ie, feeds into the gastrointestinal tract); second, when the infant has an ostomy and is receiving primarily enteral nutrition without TPN; and third, when/if the infant has a surgery to reconnect the bowel and remove the ostomy. Using stable isotope techniques for the second and third parts, we will measure intake compared to excretions (stool in ostomy and urine). A stable isotope is naturally occurring form of a mineral that we can measure, or trace, in the body. It is not radioactive and there are no known risks from it.

Part 1: This part will not include any stable isotopes. We will collect the ostomy and urine output for 24 hours to determine the zinc and copper content of the ostomy output and the urine. A small collection of blood (2 mL) will also be obtained at the same time other routine blood tests are being done. This blood will be tested for zinc, copper, and ceruloplasmin levels. If the infant has a replogle or other gastric tube, gastric residuals will be collected during the same 24 hours that stool from the ostomy is collected. If for some reason Part 1 is not able to be performed before the subject meets the criteria for Part 2, the subject will not be dropped. Part 1 will be considered optional. The following will be measured: zinc intake (from the zinc content of the TPN), endogenous fecal excretion (from the ostomy and gastric outputs) and urinary zinc excretion (from the urine collection). Zinc balance will be estimated from the difference in zinc intake and zinc output (in the ostomy, urine, and gastric fluid). Copper balance will be measured from the difference in copper intake (in TPN) and copper losses (in the ostomy, urine and gastric fluid).

Part 2: The second part of the study will occur when the infant has reached full enteral feedings (minimum of 100 cc/kg/day) and TPN has been discontinued. This part of the study will include stable isotopes. Infants should be receiving a steady state volume and concentration of feedings per kg for at least two (2) days and throughout the first 24 hours of the sample collection period. The time recorded that the infant receives the first isotope will mark the beginning of the sample collection period. Infants may be receiving either breast milk (fortified or unfortified) or infant formula. If the infant is receiving breast milk, a 10mL sample of breast milk will be obtained to determine zinc and copper content. Zinc and copper contents of infant formula will be determined from published tables by the manufacturer. The infant will receive 1 mg Zn67 and 80 mcg Cu65 stable isotope orally mixed into one of the infant's morning feedings on the study day. In addition, the infant will receive 0.1 mg Zn70 intravenous stable isotope. Stool will be collected from the ostomy bag for 72 hours. A urine bag will be placed on the infant's skin to collect all the urine for 24 hours, followed by a spot urine sample collection twice a day for three (3) days after the isotope infusion. The final urine collection should occur at approximately 96 hours after the isotope infusion. A small amount of blood (2 mL) will also be taken at the time of the intravenous isotope infusion. This blood will be tested for zinc, copper, and ceruloplasmin levels. Fractional zinc absorption and endogenous fecal zinc excretion will be measured using stable isotopes. Urinary excretion will be measured from the urine collection. Zinc balance will be calculated from the difference in absorbed zinc (intake x fractional absorption) and zinc losses (urinary excretion and endogenous fecal zinc excretion). Fractional copper absorption will be measured from the difference in intake of Cu65 and the losses of Cu65 (in the ostomy and urine). Copper balance will be measured from the difference in total copper intake and total copper losses (in the ostomy and urine).

Part 3: The third part of the study will occur after the infant has a surgery to reconnect the bowel and remove the ostomy. A spot urine sample will be obtained prior to the stable isotope infusion to ensure that isotope previously consumed/infused will not be considered in the data analysis for this part of the study. The stable isotope study will occur whenever the infant's bowel has been reconnected and the infant has achieved a steady volume and concentration of feedings per kg (minimum of 100 cc/kg/day) for at least 2 days. This volume will continue throughout the first 24 hours of the sample collection period. Infants may be receiving either breast milk (fortified or unfortified) or infant formula. If the infant is receiving breast milk, a 10mL sample of breast milk will be obtained to determine zinc and copper content. Zinc and copper contents of infant formula will be determined from published tables by the manufacturer.

As the ostomy bag has been removed, it will be difficult to obtain stool samples for 72 hours. Therefore, we will only measure zinc urine excretion, not secretion and will not be able to assess copper balance at this time point. The infant will receive 1 mg Zn67 orally mixed into one of the infant's morning feedings on the study day. In addition, the infant will receive 0.1 mg Zn70 intravenously. A small collection of blood (2 mL) will also be taken at the time of the isotope infusion. This blood will be tested for zinc, copper, and ceruloplasmin levels. One spot urine sample will be obtained at 96 hours after the first isotope is received.

Study-related information will be recorded from the medical record and will include type and volume of enteral feedings, volume and concentrations of TPN, anthropometrics, nutrition-related lab results from routine blood draws (ie, BUN, creatinine, electrolytes, bilirubin, calcium, phosphorus, alkaline phosphatase, and triglycerides), and ostomy and urine output.

Recognizing that there is the possibility that not every infant will have a surgery to reconnect the bowel, the consent form will clearly state that their child may or may not be eligible for Part 3.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ileostomy due to any disease or condition (i.e., necrotizing enterocolitis, intestinal atresias, gastroschisis, or intestinal perforations)
* Minimum birth weight of 500g
* Likely to survive

Exclusion Criteria:

* Dysmotility of the gastrointestinal system
* Major congenital anomalies, including heart disease
* Meconium ileus
* Not expected to survive for at least 2 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected from the patient population at the Neonatal Intensive Care Units of Texas Children's Hospital and Ben Taub General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Abrams, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] Wastney ME, Angelus PA, Barnes RM, Subramanian KN. Zinc absorption, distribution, excretion, and retention by healthy preterm infants. Pediatr Res. 1999 Feb;45(2):191-6. doi: 10.1203/00006450-199902000-00006. PMID 10022589
- [Background] Marriott LD, Foote KD, Kimber AC, Delves HT, Morgan JB. Zinc, copper, selenium and manganese blood levels in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2007 Nov;92(6):F494-7. doi: 10.1136/adc.2006.107755. Epub 2007 Apr 27. PMID 17468128
- [Background] Jalla S, Krebs NF, Rodden D, Hambidge KM. Zinc homeostasis in premature infants does not differ between those fed preterm formula or fortified human milk. Pediatr Res. 2004 Oct;56(4):615-20. doi: 10.1203/01.PDR.0000139428.77791.3D. Epub 2004 Aug 4. PMID 15295087
- [Background] Sandstrom B, Andersson H, Kivisto B, Sandberg AS. Apparent small intestinal absorption of nitrogen and minerals from soy and meat-protein-based diets. A study on human ileostomy subjects. J Nutr. 1986 Nov;116(11):2209-18. doi: 10.1093/jn/116.11.2209. PMID 3025388
- [Background] Woolf GM, Miller C, Kurian R, Jeejeebhoy KN. Nutritional absorption in short bowel syndrome. Evaluation of fluid, calorie, and divalent cation requirements. Dig Dis Sci. 1987 Jan;32(1):8-15. doi: 10.1007/BF01296681. PMID 3792183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the Neonatal Intensive Care Unit at Texas Children's Hospital between September 2008 and May 2010.
Groups:
- Observational Group: Infants admitted to the NICU of Texas Children's Hospital, Houston, TX who had a jejunostomy or ileostomy were recruited for the study. Neonates were enrolled if they had a jejunostomy or ileostomy and if their birth weight was > 500 grams. Infants were excluded from the study if they had any other major congenital anomalies (including congenital heart disease and cystic fibrosis), or if they were believed to be unlikely to survive to hospital discharge based on their cardiopulmonary disease.
Period: Overall Study
Arm/Group | Observational Group
Started | 17
Completed | 13
Not Completed | 4
Not completed — Death | 1
Not completed — Transfer to another facility | 2
Not completed — Discharge home prior to end of study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Observational Group
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days of life] | 44 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Zinc Absorption
Description: Zinc fractional absorption was measured using a dual tracer stable isotope method in which 67Zn was given orally with a single feed followed immediately by infusion of 70Zn intravenously. A spot urine sample was collected 96 hours after the infusion and the relative dose-corrected enrichments used to calculate fractional absorption at the time oral isotope was administered.
  Tracer:tracee ratios (TTR), measured by ICP-MS, were used to calculated fractional zinc absorption.
Time Frame: 96 hours after single feed infusion
Population: Relationships between zinc absorption, zinc excretion (urine or fecal) and zinc balance, and potential explanatory variables were analyzed using the GLM model function of JMP 7 for Macintosh (SAS inc, Cary, NC). Simple and multiple regression analysis were used as appropriate. Significance was assumed at a p < 0.05.
Measure: Mean (Standard Deviation); unit: fractional zinc absorption (%)
Arm/Group | Observational Group
Number analyzed (Participants) | 13
fractional zinc absorption (%) | 10.9 (5.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was reported annually up to 2 years.
Arm/Group | Observational Group
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
Only 10 infants achieved a majority of enteral feeds with the ostomy in place, of which only 7 were fully enterally fed at the time of the study. This is a mixed group, but nonetheless representative of infants with small intestinal ostomies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes